CLINICAL TRIAL: NCT01281982
Title: (11C)N-Desmethyl-Loperamide as a Marker of P-Glycoprotein Function in Patients With Gliomas
Brief Title: (11C)dLop as a Marker of P-Glycoprotein Function in Patients With Gliomas
Status: Terminated | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110081; 11-C-0081
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2012-09-24

CONDITIONS: Low Grade Glioma; Glioblastoma Multiforme; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Oligoastrocytoma
Keywords: Imaging; Gliomas; Pet Scan; Blood Brain Barrier; P-Glycoprotein; Brain Tumor; Glioma; Glioblastoma Multiforme; Astrocytoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Brain Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- The blood-brain barrier helps to protect the central nervous system (brain and spinal cord) from harmful toxins, but also prevents potentially useful chemotherapy from reaching brain tumors. The barrier is formed by tight connections between blood vessel cells and molecules found on the surface of brain blood vessels such as Permeability-glycoprotein (Pgp). Pgp may influence whether patients with brain tumors known as gliomas respond to chemotherapy and what side effects they may experience. The compound (11C)N-desmethyl-loperamide ((11C)dLop) reacts to Pgp molecules, and therefore may be used with positron emission tomography (PET) imaging to study the blood brain barrier.

Objectives:

- To study the ability of PET imaging with (11C)dLop to evaluate the blood brain barrier in brain tumor patients.

Eligibility:

- Individuals at least 18 years of age who have a brain tumor with characteristics that may be imaged with techniques such as magnetic resonance imaging (MRI) andPET.

Design:

* Participants will be screened with a full physical examination and medical history, blood and urine tests, and tumor imaging studies (fluorodeoxyglucose PET and MRI scans with contrast agent).
* The (11C)dLop scan will take 1 hour to perform. Participants will be asked to return for blood and urine tests approximately 24 hours after the PET scan.
* Participants will have followup visits at least every 4 months by repeating a complete history and physical exam and brain MRI. Participants may have repeat scans with (11C)dLop at various points in the course of cancer treatment, but will not have these scans more than twice in a 12-month period.
* Participants will be followed for as long as possible during treatment to see if imaging with (11C)dLop correlates with response to the treatments.

DETAILED DESCRIPTION:
BACKGROUND:

A potential impedance to successful glioma chemotherapy is sanctuary for tumor behind the blood brain barrier. P-glycoprotein (Pgp) is an efflux transporter encoded by MDR1 that contributes to the functional regulation of substrates across the cerebrovasular endothelium. Pgp activity in patients with gliomas may influence response to therapy and neurotoxicity. (11C) N-desmethyl-loperamide (11C)dLop) is a radioligand substrate for Pgp, and PET imaging with this molecular marker may provide a non-invasive, in vivo method of examining Pgp function in brain tumor patients.

OBJECTIVES:

Primary:

-To measure the uptake of (11C)N-desmethyl-loperamide ((11C)dLop) using PET imaging as a marker of Pglycoprotein function in patients with intracranial gliomas

Secondary:

* Correlate (11C)dLop PET uptake with perfusion MRI parameters and FDG PET uptake for volumes of interest (VOI) determined by the baseline MRI
* Develop exploratory data for the correlation of (11C)dLop PET imaging with patient outcomes such as response to therapy, survival, and neurotoxicity
* Develop exploratory data for the correlation of (11C)dLop PET imaging with immunohistochemical and molecular genomic assays of MDR1 and Pgp

ELIGIBILITY:

Patients with predominantly non-enhancing intracranial gliomas will be eligible.

DESIGN:

This is a pilot study of (11C)dLop PET imaging in 10 patients with intracranial glioma. Standard uptake values (SUVs) corrected for cerebral blood flow determined by (15O)H20 PET scans will be correlated to DCE-MRI (obtained within prior 2 weeks) and FDG-PET (obtained within prior 4 weeks) to characterize locoregional differences in Pgp function. When available, correlative studies performed on archived tumor tissue acquired immediately subsequent to (11C)dLop scanning will include immunohistochemical assays of Pgp expression, as well as characterization of MDR1 polymorphisms. Patient case histories will be followed longitudinally to make observations about how (11C)dLop imaging may correlate with patient outcomes such as response to therapy, survival, and neurotoxicity.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with histologically proven intracranial glioma will be eligible for this protocol. Eligible histologies include glioblastoma multiforme (GBM), gliosarcoma (GS), anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), malignant astrocytoma NOS (not otherwise specified), low grade astrocytoma (LGA), low grade oligoastocytoma (LOA), and low grade oligodendroglioma (LGO). Patients with radiographically diagnosed or suspected low grade glioma will also be eligible.
* Patients having undergone recent resection will be eligible as long as all of the following conditions apply:

  * They have recovered from the effects of surgery, not to have been performed within 2 weeks of the study scan.
  * Residual enhancing or non-enhancing disease following resection of recurrent tumor is mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a CT/ MRI should be done:
  * no later than 96 hours in the immediate post-operative period, or
  * at least 4 weeks post-operatively, and
  * within 14 days of registration, and
  * on a steroid dosage that has been stable for at least 5 days.
* Normal organ and marrow function defined as: total leukocyte count greater than or equal to 3000 cells/ul, ANC greater than or equal to 1500 cells/ul, platelet count greater than or equal to 100,000 cells/ul, serum creatinine less than or equal to 2.0 X upper limit of normal, and bilirubin less than or equal to 1.5X upper limit of normal, hemoglobin greater than or equal to 9.0 g/dL , serum calcium less than12.0 mg/dL, AST/ALT less than or equal to1.5 times the upper limit of normal, PT less than or equal to1.5 ULN.
* All patients or their previously designated DPA (if the patient is deemed by the treating physician to be impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) must sign an informed consent indicating that they are aware of the investigational nature of this study.
* Patients must be greater than or equal to 18 years old.
* Patients must have a Karnofsky performance status of greater than or equal to 60.
* Patients must not have any significant medical illnesses that in the investigator s opinion cannot be adequately controlled with appropriate therapy or would compromise the patients ability to tolerate this study.
* This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race. Minorities will actively be recruited to participate.

EXCLUSION CRITERIA:

* Patients who, in the view of the treating physician, have significant active cardiac, hepatic, renal, or psychiatric diseases are ineligible.
* Patients who have an active infection.
* Pregnant (positive pregnancy test) or nursing women.
* Patients cannot take loperamide within three days of (11C)dLop imaging.
* Concurrent use of a Pgp inducer as listed in Appendix A within 2 weeks of a study scan. Use of these medications is allowed over the course of participation in the study, but must not be administered within 2 weeks of the study imaging.
* Prior participation in other research protocols or clinical care in the last year such that radiation exposure, including that from this protocol, would exceed the guidelines set by the Radiation Safety Committee (RSC).
* Patients who have any contraindication to gadolinium enhanced MRI.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-01-13; Study Completion 2012-09-24

CONTACTS AND LOCATIONS:
Overall Officials: Teri N Kreisl, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hochberg FH, Pruitt A. Assumptions in the radiotherapy of glioblastoma. Neurology. 1980 Sep;30(9):907-11. doi: 10.1212/wnl.30.9.907. PMID 6252514
- [Background] Bloom HJ. Combined modality therapy for intracranial tumors. Cancer. 1975 Jan;35(1):111-20. doi: 10.1002/1097-0142(197501)35:13.0.co;2-#. PMID 162849
- [Background] Salazar OM, Rubin P, McDonald JV, Feldstein ML. High dose radiation therapy in the treatment of glioblastoma multiforme: a preliminary report. Int J Radiat Oncol Biol Phys. 1976 Jul-Aug;1(7-8):717-27. doi: 10.1016/0360-3016(76)90155-3. No abstract available. PMID 185174